CLINICAL TRIAL: NCT06908798
Title: The Accuracy of Fecal Calprotectin in Detecting Esophageal Varices in Egyptian Patients With Liver Cirrhosis
Brief Title: Fecal Calprotectin for Prediction of Esophageal Varices in Cirrhotic Patients
Status: Recruiting | Type: Observational
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Rania Mamdouh Elkafoury, Lecturer of Tropical Medicine, Tanta University
Other Study IDs: 36264PR983/12/24
Record Dates: First submitted 2025-03-27; First posted 2025-04-03 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Esophageal Varices
Keywords: Fecal calprotectin; esophageal varices; liver cirrhosis
MeSH Terms: conditions — Esophageal and Gastric Varices; Liver Cirrhosis

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- cirrhotic patients with esophageal varices: 52 cirrhotic patients with esophageal varices.
  Interventions: Diagnostic Test: fecal calprotectin
- cirrhotic patients without esophageal varices: 52 cirrhotic patients without esophageal varices.
  Interventions: Diagnostic Test: fecal calprotectin
- control group: 52 healthy subjects as a control.
  Interventions: Diagnostic Test: fecal calprotectin

INTERVENTIONS:
Diagnostic Test: fecal calprotectin — fecal calprotectin test measures calprotectin protein in a stool sample. fecal calprotectin acts as a surrogate for gastrointestinal inflammation (e.g., inflammatory bowel disease, infectious gastroenteritis, acute appendicitis, peptic ulcer disease, coeliac disease, non-steroidal anti-inflammatory drugs (NSAID)-induced enteropathy)

SUMMARY:
The goal of this cross-sectional observational study is to evaluate the accuracy of fecal calprotectin versus non-invasive scores in assessing the presence and grading of esophageal varices in Egyptian patients.

Researchers will compare fecal calprotectin levels in cirrhotic patients with and without esophageal varices (EVs) and healthy subjects. researchers will also evaluate the performance of fecal calprotectin, AST to platelet ratio index (APRI) score, fibrosis-4 (FIB-4) score, albumin-bilirubin (ALBI) score, platelet-albumin-bilirubin (PALBI) score, and platelet-spleen diameter ratio (PSR) for predicting esophageal varices.

Participants will undergo history-taking, clinical examination, laboratory investigations, fecal calprotectin, abdominal ultrasonography, and upper endoscopy. Endoscopic grading of esophageal varices will be done using Paquet's classification. The APRI, FIB-4, ALBI, PALBI, and PSR scores will be calculated. The performance of fecal calprotectin for predicting EVs will be compared versus other non-invasive scores.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Liver cirrhosis

Exclusion Criteria:

* Patients aged < 18 years.
* Inflammatory bowel disease.
* Infectious gastroenteritis.
* Malignancy.
* Patients on proton pump inhibitors or NSAID.
* Patients with spontaneous bacterial peritonitis.
* Patients with hepatic encephalopathy.
* Unwilling to participate in our study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This cross-sectional observational study will be carried out on 156 patients who will be enrolled from the endoscopy unit in the Tropical Medicine and Infectious Diseases Department, Tanta University Hospital, Egypt. The start of research will begin in December 2024 and will end in December 2025.
Sampling Method: Probability Sample
Enrollment: 156 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
measuring fecal calprotectin level (microgram/gram) for predicting esophageal varices | through study completion, an average of 1 year

SECONDARY OUTCOMES:
comparing fecal calprotectin versus non-invasive scores for predicting esophageal varices | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Rania M Elkafoury, MD, Principal Investigator — Tropical medicine and infectious diseases Department, Faculty of Medicine, Tanta University
Locations (1):
- Tanta University Hospitals, Tanta, Gharbyea, Egypt